CLINICAL TRIAL: NCT01075893
Title: Changes in Stem Cells of the Colon in Response to Increased Risk of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: McCallum-001
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2016-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Stem cells; Ulcerative colitis; Polyps
MeSH Terms: conditions — Colorectal Neoplasms; Colitis, Ulcerative; Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rectal pinch biopsies - x 9 (10 cm from anal verge)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adenomatous polyp: Patients who have begun the polyp-cancer sequence (ie. are in polyp surveillance after excision of a prior adenomatous polyp) will be used to test those patients at higher risk of colorectal.
- Patients at normal risk of cancer: Patients found to have endoscopically and histological normal mucosa.
- Ulcerative colitis: Patients who are under surveillance for known ulcerative colitis will be used to test those patients at higher risk of colorectal.

SUMMARY:
Colorectal cancer is a common disease worldwide. Increasing evidence is demonstrating that colorectal cancers arise from 'cancer stem cells.' Stem cells in the colon reside at the bottom of thousands of microscopic crypts throughout the wall of the colon. They create all the cells lining the bowel wall. These cells are created in the base of the crypt and ascend to the top acquiring the characteristics of mature cells of the bowel wall as they ascend.

It is now thought that colorectal cancer cells arise from stem cells where the genetic material regulating growth and division of the stem cell has become defective. This leads to unregulated production of cells which in turn have defective genetic information and cancer formation.

Prior studies have demonstrated that the earliest changes before a cancer develops are changes in cellular proliferation. Now that reliable markers to identify stem cells have been found, the researchers aim to investigate stem cell numbers and changes in distribution in those at normal risk of colorectal cancer and those at higher risk. The researchers hypothesise that changes in cellular proliferation at the top of the crypt in individuals at higher risk of colorectal cancer are due to a change in the number of stem cells in the crypt base.

ELIGIBILITY:
Inclusion Criteria:

* Referred for endoscopy at participating centre

Exclusion Criteria:

* Age <16 or >85
* Familial polyposis syndrome
* Lynch syndrome
* Known colorectal tumour
* Previous colorectal resection
* Pregnancy
* Chemotherapy in last 6 months
* Therapy with aspirin/other nonsteroidal anti-inflammatory drug (NSAID)
* Other immunosuppressive medication
* Incomplete left sided examination
* Colorectal carcinoma found at endoscopy
* Iatrogenic perforation at endoscopy
* Colorectal cancer on histology
* Microscopic colitis on histology

For the colitis group

* Simple clinical colitis activity index (SCCAI) score > 5

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred for lower gastrointestinal (GI) endoscopy at a participating centre will be considered for inclusion. Patients with a previous adenomatous polyp resection under surveillance will be considered for inclusion to the polyp group. Patients with ulcerative colitis under surveillance will be considered for inclusion to the ulcerative colitis group.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of stem cells in the colonic crypt | On day of endoscopy

SECONDARY OUTCOMES:
Stem cell position in colonic crypt | On day of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Iain JD McCallum, MBChB MRCS, Principal Investigator — Newcastle University, UK; John C Mathers, PhD, Study Chair — Newcastle University, UK; Seamus B Kelly, MD FRCS, Study Director — Newcastle University, UK; Mike Bradburn, MD FRCS, Study Director — Northumbria NHS foundation trust
Locations (2):
- United Kingdom (2):
  - Wansbeck General Hospital, Ashington, Tyne & Wear
  - North Tyneside Hospital, North Shields, Tyne & Wear

REFERENCES:
- [Background] Dronamraju SS, Coxhead JM, Kelly SB, Burn J, Mathers JC. Cell kinetics and gene expression changes in colorectal cancer patients given resistant starch: a randomised controlled trial. Gut. 2009 Mar;58(3):413-20. doi: 10.1136/gut.2008.162933. Epub 2008 Oct 31. PMID 18978177
- [Background] Barker N, van Es JH, Kuipers J, Kujala P, van den Born M, Cozijnsen M, Haegebarth A, Korving J, Begthel H, Peters PJ, Clevers H. Identification of stem cells in small intestine and colon by marker gene Lgr5. Nature. 2007 Oct 25;449(7165):1003-7. doi: 10.1038/nature06196. Epub 2007 Oct 14. PMID 17934449